CLINICAL TRIAL: NCT06761690
Title: Hybrid Simulation Training on Nursing Students' Wound Care Knowledge, Skills, and Compassion Competence: A Randomized Controlled Trial
Brief Title: Hybrid Simulation Training on Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EDA UNAL (Other)
Responsible Party: Sponsor-Investigator, EDA UNAL, Assoc. Prof. Dr., Uludag University
Organization: Uludag University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: BursaUludagUEda
Record Dates: First submitted 2024-12-07; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Wounds; Wounds and Injuries; Wound Heal
Keywords: wound care, nursing student, simulation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: A randomized controlled study was conducted. The experimental group received hybrid simulation wound care training. The control group received theoretical training and additional materials to perform wound dressing, just like all students.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Hybrid simulated wound training
  Interventions: Other: hybrid simulated wound training
- Control (No Intervention): Received standard education

INTERVENTIONS:
Other: hybrid simulated wound training — hybrid simulated wound training
  Arms: experimental

SUMMARY:
To investigate the effects of hybrid simulation training on nursing students' wound care knowledge, skills and compassion competence.

Design: This study was a randomised controlled experimental design. Methods: The study comprised nursing students divided into two groups: the experimental group (n=42) and the control group (n=38). All participants received a two-class-hour (100 minutes) training session covering skin anatomy, wound formation, wound characteristics, wound types, appropriate dressing selection, and compassion in nursing.

Nursing students' wound care knowledge was assessed using a knowledge test, while their skills in wound physical assessment, intervention, and dressing application were evaluated through a structured objective clinical examination.

Additionally, students' compassion competencies were measured using the Compassion Competency Scale.

DETAILED DESCRIPTION:
Wounds are divided into acute and chronic Acute wounds, characterized by their sudden appearance on the skin, include various types such as surgical wounds, traumatic wounds, and burn wounds Inadequate care of acute wounds leads to their transformation into chronic wounds. Nurses and nursing students have low levels of wound management competence Compassion is defined as an internal emotion that motivates individuals to relieve the suffering of others. Compassionate care can be formally defined as the recognition and understanding of an individual's suffering, characterized by deep empathy and understanding.

Provides a safe environment for nursing students to solve and develop critical attitudes. In hybrid simulation, the use of wound attachments and wound moulages facilitates accurate wound identification, classification, appropriate intervention, and correct wound dressing. The development of compassion competence through simulation training to improve nursing students' knowledge and skills in wound care has not yet been examined. The purpose of this study was to investigate the effects of hybrid simulation training on nursing students' wound care knowledge, wound assessment and dressing skills, and compassion competence.

Methods This study was a randomized controlled experimental study conducted with nursing students. The study consisted of nursing students divided into two groups: experimental group (EG) (n=42) and control group (CG) (n=38).

This study was conducted with 3rd year nursing students (n=155) enrolled in a four-year undergraduate nursing program at Bursa Uludağ University, and they were invited to participate in this research in the spring semester of the 2023-2024 academic year.

Participants who were transitioning to internship practice, had no previous experience with simulation training, and wound care training were included.

Theoretical Training Sessions All students received training on acute and chronic wounds. Detailed explanations were provided through case scenarios and visual videos. After the theoretical training, students were given information and skills were assessed with a knowledge test and structured clinical exam. The control group received theoretical training and applied wound dressings on additional parts.

Students were given simulation training. A patient who had a traffic accident resulting in open and closed wounds of different degrees, sizes and depths on the chest, right hand and arm a scenario was developed that includes.

ELIGIBILITY:
Inclusion Criteria:

* Third year nursing student
* First to attend simulation training

Exclusion Criteria:

* Not a third year nursing student
* Have attended simulation training before

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Wound information ( min=0, Mak=20 points) | 2 week
  survey
Wound skill ( min=0, Mak=42 points) | 2 week
  survey
Compassion Competence Scale (min=1 Mak=5 points) | 2 week
  Compassion Competence Scale

CONTACTS AND LOCATIONS:
Overall Officials: Betül SANLAN, Study Chair — Medical Sciences, University of Surrey
Locations (2):
- Turkey (Türkiye) (2):
  - Bursa Uludag University, Bursa, Nilüfer
  - Uludag Üniversty, Bursa

IPD SHARING:
Plan to Share IPD: No
The study was published before the study was published